CLINICAL TRIAL: NCT07362043
Title: Assessment of a Hand-held Femtosecond Laser to Perform Anterior Capsulorhexis During Cataract Surgery (Post-market Study)
Acronym: PMCF_SEQ_Rx
Status: Recruiting | Type: Observational
Sponsor: Helix Surgical (Industry)
Collaborators: Santé Atlantique - Saint-Herblain - France (Unknown)
Responsible Party: Sponsor
Other Study IDs: CER-BDX 2025-157
Record Dates: First submitted 2026-01-05; First posted 2026-01-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cataract Surgery
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cataract surgery with Rx, a handheld femtosecond laser for anterior capsulotomy (CE-marked device used as intended) — Cataract surgery with Rx, a handheld femtosecond laser for anterior capsulotomy

SUMMARY:
The goal of this observationnal study is to supplement the data collected in the pre-market study and confirm the rate of capsular ruptures due to Rx (reducing its related confidence interval).

During cataract surgery, an artificial lens is placed into the capsular bag. The main question this study aims to answer is :

Is Rx use associated with a rate of caspular ruptures lower than 2% ? Medical records of participants having cataract surgery with Rx laser as part of their regular medical care will be assessed in order to answer the study objective.

DETAILED DESCRIPTION:
This study is a PMCF, sequential, non-interventional, prospective (follow-up: 30 ± 15 days), single-arm, single center, open trial.

Note: The design of this study is identical to the one of the Rx pre-market investigation (same design, same endpoints, same investigation site, same follow-up).

78 patients have been included in the pre-market investigation and will be used as part of dataset of the current PMCF study.

Sample size calculation (Wilson Method):

Considering the design of this study is identical to the one of the Rx pre-market investigation and that 78 patients have already been included in that pre-market clinical investigation (NCT05141370);

Assuming a rate of capsule-ruptures due to Rx < 2%;

And an upper limit ≤ 3.5%;

The maximum number of patients to be included will be 446 patients (considering 78 patients have already been included, 368 remain to be included), corresponding to 8 capsular ruptures and a rate of 1.79% with an interval of [0.91% ;3.5%].

The investigator proposes to conduct a sequential study in which the number of patients depends on a success criterion and a failure criterion as detailed below.

As the study is sequential, interim analyses at the end of each sequence are planned to examine whether the objective of an upper limit of rupture rate ≤3.5% (success) is achieved, or whether the rupture rate equals or exceeds 2% (failure).

The study stops as soon as a success or failure criterion is verified.

Sequence 1:

- 106 patients to reach:

* Success: 0 capsular rupture -> superior limit ≤ 3.5%
* Failure: ≥ 3 capsular ruptures -> a rupture rate ≥ 2%

If 1 ≤ number of capsular ruptures ≤2 the trial continues

Sequence 2:

- 158 patients to reach:

* Success: 1 capsular rupture -> superior limit ≤ 3.5%
* Failure: ≥ 4 capsular ruptures -> a rupture rate ≥ 2%

If 2 ≤ number of capsular ruptures ≤3 the trial continues

Sequence 3:

- 205 patients to reach:

* Success: 2 capsular ruptures -> superior limit ≤ 3.5%
* Failure: ≥ 5 capsular ruptures -> a rupture rate ≥ 2%

If 3 ≤ number of capsular ruptures ≤4 the trial continues

Sequence 4:

* 248 patients to reach:

  * Success: 3 capsular ruptures -> superior limit ≤ 3.5%
  * Failure: ≥ 5 capsular ruptures -> a rupture rate ≥ 2%

If 4 capsular ruptures the trial continues

Sequence 5:

- 290 patients to reach:

* Success: 4 capsular ruptures -> superior limit ≤ 3.5%
* Failure: ≥ 6 capsular ruptures -> a rupture rate ≥ 2%

If 5 capsular ruptures the trial continues

Sequence 6:

- 330 patients to reach:

* Success: 5 capsular ruptures -> superior limit ≤ 3.5%
* Failure: ≥ 7 capsular ruptures -> a rupture rate ≥ 2%

If 6 capsular ruptures the trial continues

Sequence 7:

- 370 patients to reach:

* Success: 6 capsular ruptures -> superior limit ≤ 3.5%
* Failure: ≥ 8 capsular ruptures -> a rupture rate ≥ 2%

If 7 capsular ruptures the trial continues

Sequence 8:

- 408 patients to reach:

* Success: 7 capsular ruptures -> superior limit ≤ 3.5%
* Failure: ≥ 9 capsular ruptures -> a rupture rate ≥ 2%

If 8 capsular ruptures the trial continues

Sequence 9:

* 446 patients to reach:

  * Success: 8 capsular ruptures -> superior limit ≤ 3.5%
  * Failure: ≥ 9 capsular ruptures -> a rupture rate ≥ 2%

    446 patients is the maximum number of patients to be included in the study, as no condition other than success or failure can be verified.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years);
* Diagnosed with cataract requiring surgery according to current guidelines;
* Eligible to lens removal by phacoemulsification and replacement by a prosthetic lens under local anesthesia;
* Who confirmed their non-opposition to data collection

Exclusion Criteria:

* Patient already operated with Rx for the first eye.
* Any contra-indication to cataract surgery;
* Patients with an ACD (Anterior Chamber Depth) less than 1.8mm and greater than 4.2mm;
* Corneal disease or pathology that prevents corneal applanation or that may interfere with or hinder laser beam transmission;
* Presence of blood or any other element that hinders the propagation of light between the epithelium and the anterior surface of the lens where the capsulotomy will be performed;
* Weak pupil dilation or severely off-center pupil that prevents the iris from retracting adequately to the periphery (dilations < 6.5mm in diameter are excluded);
* Abnormal tilt of the lens (> 7 degrees) ;
* Significant preoperative ocular hypotonia or hypertonia;
* Presence of an intra-corneal implant;
* Active or unstabilized ocular surface disease including abnormal corneas (e.g., epithelial dystrophies,recurrent ulcers, infectious foci, conjunctivitis, severe dry syndromes);
* History of lens disease or zonular instability;
* Any perforating incision of the eyeball that may result in leakage during corneal applanation;
* Presence of a limbal tumor obstacle that may interfere with stabilization of the device on the limbus: pterygium, limbal tumor, filter bubble, etc.
* Patients under guardianship, trusteeship or deprived of liberty;
* Patients unable to give their non-opposition for data collection for psychiatric, cognitive or linguistic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients eligible for cataract surgery
Sampling Method: Probability Sample
Enrollment: 446 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Rate of capsule-ruptures due to Rx | During surgery
  The investigator considers a rupture of the capsule will be Rx-related if:
  * There are peripheric tears that can generate the rupture of the capsule during or at the end of rhexis removal;
  * AND these tears generate the rupture of the capsule during surgery.

SECONDARY OUTCOMES:
Continuity of the capsulorhexis (success / failure) | During surgery
  Success is achieved if:
  * the anterior capsule is completely cut (rhexis is free floating or easy to remove)
  * AND there are no peripheric tears that can generate the rupture of the capsule at the end of rhexis removal.
Adverse device effects | During surgery, 4 days after surgery (4 ± 2 days), 30 days after surgery (30 ± 15 days)
  Collection of adverse device effects by the investigator on the retina, on the cornea, on the posterior capsula and other adverse device effects

OTHER OUTCOMES:
Patient's perception about Rx use (exploratory endpoint) | During surgery
  Patient's rating, on a 4-degree-scale of discomfort, and overall satisfaction with the use of Rx
Rx usability (exploratory endpoint) | During surgery
  o Investigator's rating, on a 4-degree-scale of several surgical steps: preparing the device before surgery; handling the device in the operating field; visualizing the eye through the device; centering the device on the capsule; keeping the device in the correct position; activating the laser beam; removing the device from the eye after capsulorhexis, etc.
  o Measure of laser power delivered by Rx before each surgery.
Circularity of the capsulorhexis (exploratory endpoint) | During surgery
  Ratio : real capsulorhexis surface in mm2 / intended capsulorhexis surface in mm2
Distance between the center of the rhexis and the center of the pupil / iris (in mm) (exploratory endpoint) | During surgery
Visual acuity by refractometry and its change from baseline to 30 days after surgery (exploratory endpoint) | During surgery, 4 days after surgery (4 ± 2 days), 30 days after surgery (30 ± 15 days)
Difference in between expected post-operative visual acuity and real post-operative visual acuity (exploratory endpoint) | 30 days after surgery (30 ± 15 days)
Successful placement of the IOL into the capsular bag (success/failure) (exploratory endpoint) | During surgery, 4 days after surgery (4 ± 2 days), 30 days after surgery (30 ± 15 days)
  Qualitative evaluation by the investigator/surgeon based on its surgeon expertise
Intraocular pressure and its evolution form baseline to 30 days after surgery (exploratory endpoint) | During surgery, 4 days after surgery (4 ± 2 days), 30 days after surgery (30 ± 15 days)
Corneal thickness and its evolution from baseline to 30 days after surgery (exploratory endpoint) | During surgery, 4 days after surgery (4 ± 2 days), 30 days after surgery (30 ± 15 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Santé Atlantique, Saint-Herblain, France